CLINICAL TRIAL: NCT00821665
Title: Blood Glucose Homeostasis in Type 2 Diabetes: the Effects of Saccharose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Suikerstichting Nederland (Baarn) (Unknown)
Responsible Party: Dr. L.J.C. van Loon Ph.D, Maastricht University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 07-3-004
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Type 2 Diabetes; Glycemic Control
Keywords: Type 2 diabetes; Glycemic control; (postprandial) Hyperglycemia; Sucrose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose (Experimental): Sucrose
  Interventions: Dietary Supplement: Sucrose consumption
- Water (Placebo Comparator): Water
  Interventions: Dietary Supplement: water consumption

INTERVENTIONS:
Dietary Supplement: Sucrose consumption — Sucrose
  Arms: Sucrose
Dietary Supplement: water consumption — water
  Arms: Water

SUMMARY:
Hyperglycemia forms a direct and independent risk factor for the development of cardiovascular co-morbidities in type 2 diabetes. Consumption of sucrose-sweetened soft drinks might further increase the prevalence of hyperglycemic episodes.

The objective of the study was to assess glycemic control in type 2 diabetes patients and healthy lean and obese controls under strict dietary standardization but otherwise free living conditions, with and without the consumption of soft drinks.

ELIGIBILITY:
Inclusion Criteria:

Lean NGT Group

* Normoglycemic (according to 2006 ADA guidelines)
* BMI < 27 kg/m2

Obese NGT Group

* Normoglycemic
* BMI 30- 35 kg/m2

Obese type 2 diabetes Group

* BMI 30- 35 kg/m2
* Oral blood glucose lowering medication

Exclusion Criteria:

* Exogenous insulin use
* Cardiac disease (any cardiac event in the last 5 years)
* HbA1c >10%
* Microalbuminuria: albumin:creatinine ratio >2,5

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Hyperglycemia | 24h

SECONDARY OUTCOMES:
Hyperglycemia | Postprandially

CONTACTS AND LOCATIONS:
Overall Officials: Luc J van Loon, Ph.D, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limbrug, Netherlands